CLINICAL TRIAL: NCT06200480
Title: Nurse Intervention Trial: The Evaluation of Usefulness of a Headache Nurse
Brief Title: Nurse Intervention Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Haukeland University Hospital (Other); Oslo University Hospital (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-554940
Record Dates: First submitted 2023-12-14; First posted 2024-01-11 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Migraine; Chronic Tension-Type Headache; Cluster Headache; Hemicrania Continua
MeSH Terms: conditions — Migraine Disorders; Cluster Headache

STUDY DESIGN:
Intervention Model Description: Open-label randomized prospetive study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone by nurse (Active Comparator): The headache patients will be contacted by nurse by phone after approximately 2 week and 6 week after start of preventive medical treatment. The patient will have a follow-up visit by neurologist after 3 months.
  Interventions: Other: Telephone by nurse
- Patient-initiated follow-up (No Intervention): The headache patient contact their general practitioner (GP) and/or the neurologist by a study-specific email if they have questions regarding the preventive medical treatment

INTERVENTIONS:
Other: Telephone by nurse — Patient-initiated follow-up at week 2 and 6
  Arms: Telephone by nurse

SUMMARY:
This randomized open-label prospective study focus on headache patients initiating preventive treatment, where the treating physician identifies a need for follow-up visits in specialized healthcare. The study will clarify whether the implementation (compliance) and overall satisfaction of the patient are better with follow-up by a headache nurse compared to standard follow-up. Patients with signed written consent will be randomised to either group a: Telephone calls from nurse after two and 6 week or B. Patient-initiated follow-up by their general practitioner.

DETAILED DESCRIPTION:
Potential patients suitable for this study must have undergone a regular consultation with a neurologist before. This consultation includes neurological and somatic examinations, diagnosis of the type of headache based on medical history, review of a completed headache diary, and any additional conducted examinations. The consultation will also involve an assessment of the possible initiation of preventive treatment. A selection of these patients will be prescribed electronic prescriptions for at least one previously untried type of preventive medication. During the consultation, patients will receive oral and written information about the dosage and expected possible side effects of the preventive medication. Those eligible for beta-blocker initiation will undergo an electrocardiogram (EKG) after the consultation. After completing the consultation, eligible patients will receive written and oral information about the study.

Those who provide consent to participate will, during subsequent registration with the secretaries at the neurological outpatient clinic immediately after the consultation, be randomized to one of two follow-up options (A or B) for further monitoring in the coming months until the scheduled follow-up, set at approximately 3 months, or later if there is a shortage of available appointments.

Group A will be followed up by a headache nurse through telephone consultations on at least two occasions shortly after the initiation of preventive medicine. Participants in this group will be invited to a planned final follow-up appointment after approximately 3 months with a neurologist.

Group B will have patient-managed follow-up with a planned final follow-up appointment after approximately 3 months. Participants will pick up the prescribed medication and contact their general practitioner or the neurological outpatient clinic by a study-specific email if they need advice from a neurologist.

ELIGIBILITY:
Inclusion Criteria:

* One of the following headache diagnoses based on the International Classification of Headache Disorders, third edition (ICDH3): G44.2 Chronic tension-type headache and/or G43 Episodic and chronic migraine, G44.0 Episodic and chronic cluster headache, G44.8 Hemicrania Continua
* Indication for preventive medication where there is at least one alternative with the need for follow-up assessment of effectiveness.

Exclusion Criteria:

* Uncertain headache diagnosis.
* Need further investigation after the initial consultation.
* Lack of understanding of information provided in Norwegian, both verbally and in writing.
* Inability to keep a digital headache diary.
* Need treatment of other comorbid conditions requiring follow-up in specialized healthcare.
* Treatment with Onabotulinumtoxin A or Calcitonin-gene-related Peptide (CGRP) inhibitors given with three months intervals

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Compliance | 2 months
  number of participants who have carried out the prescribed preventive treatment, as in minimum duration of two months after the initial visit

SECONDARY OUTCOMES:
Number of days to at least a 30% reduction | 3 months
  Number of days from inclusion to at least a 30% reduction erate to severe headache compared to in the frequency in the last month before the initial consultation
Responders | 3 months
  Numbers of responders defined as> 50% decrease in headache days compared to in the frequency in the last month before the initial consultation

CONTACTS AND LOCATIONS:
Overall Officials: Geir Braathen, Study Chair — St. Olavs Hospital, Trondheim, Norway
Locations (1):
- St. Olavs Hospital HF, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
Publication by home page of NorHead
Supporting Information: Study Protocol, SAP, ICF
Time Frame: In the near future
Access Criteria: https://www.ntnu.no/norhead/om
URL: https://www.ntnu.no/norhead/om

REFERENCES:
- See also: Information by request — https://www.ntnu.no/norhead/om
- Available data/document: Study Protocol: NorHead — https://www.ntnu.no/norhead/om — English Study protocol available by request to the Norwegian Centre of Headache Research (NorHead)
- Available data/document: Statistical Analysis Plan: NorHead — https://www.ntnu.no/norhead/om — English SAP available by request to the the Norwegian Centre of Headache Research (NorHead)

DOCUMENTS (2):
  • Study Protocol (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT06200480/Prot_000.pdf
  • Informed Consent Form (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT06200480/ICF_001.pdf